CLINICAL TRIAL: NCT01405729
Title: Medial Patellofemoral Ligament Reconstruction: A Review of Technique, Accuracy, and Outcome
Acronym: MPFL
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Robert Burks, M.D., University of Utah
Other Study IDs: 39977
Record Dates: First submitted 2011-07-27; First posted 2011-07-29 (Estimated); Last update posted 2014-02-14 (Estimated); Status verified 2014-02

CONDITIONS: Healthy; Medial Patellofemoral Ligament Reconstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this retrospective study was to determine the accuracy of femoral tunnel placement utilizing Redfern et al's radiographic method for anatomic femoral attachment during MPFL reconstruction in addition to the resultant outcome.

DETAILED DESCRIPTION:
Reconstruction of the medial patellofemoral ligament (MPFL) has been shown to be an effective treatment for recurrent patellar instability, There has been some concern in the literature about the accuracy of femoral tunnel placement and the effect that it might have on patient outcomes.

The investigators evaluated the accuracy of MPFL placement using an intraopetative fluoroscopy technique and to assess subsequent patient outcomes.

All patients undergoing MPFL reconstruction using an intraoperative fluoroscopically guided technique between 2005 and 2010 were identified. A retrospective review of their charts and radiographs were performed and the subjects were brought back for a follow up exam, radiographic series, and Kujala questionaire.

ELIGIBILITY:
Inclusion Criteria:

* Patients having undergone the MPFL procedure, starting January 1, 2005 through February 3, 2010
* Minimum follow up of 24 months

Exclusion Criteria:

* Pregnant women
* Under 18 years of age
* Previously undergone prior MPFL surgery
* Participated in any previous research studies involving the use of ionizing radiation (either radioisotopes or diagnostic x-rays during the past 12 months.
* The participant should not volunteer for other research studies involving the use of ionizing radiation within 12 months of completing the current study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A single surgeon experience beginning in 2005 with patient's undergoing MPFL reconstruction using intra-operative fluoroscopy for proper placement of the femoral tunnel.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2010-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Radiograph measurements | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Robert T Burks, MD, Principal Investigator — University of Utah Orthopaedic Center
Locations (1):
- University of Utah Orthopedics Center, Salt Lake City, Utah, United States